CLINICAL TRIAL: NCT00002182
Title: Megestrol Acetate For Failure To Thrive In Pediatric HIV
Brief Title: A Study of Megestrol Acetate in HIV-Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamma Project - ACTU (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 266A; Gamma 005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: Placebos; Appetite Stimulants; Megestrol Acetate; Failure to Thrive
MeSH Terms: conditions — HIV Infections; Failure to Thrive | interventions — Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol acetate

SUMMARY:
The purpose of this study is to see if megestrol acetate is safe and effective in treating HIV-infected children with failure to thrive (FTT).

DETAILED DESCRIPTION:
The study design is randomized, double-blind, placebo-controlled for 12 weeks with open-label drug offered after week 12.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* Failure to thrive as defined by:
* crossing 2 percentile lines on standard weight for age curves over time or less than 5% percentile weight for age and falling from the curve or loss of 10% of baseline body weight.
* Resistant to oral nutritional supplementation (i.e., FTT despite a minimum 1-month trial of high-calorie oral supplements).
* Free of significant acute illness (mild upper respiratory tract infections allowed).
* Patients with chronic diarrhea allowed provided malabsorption and gastrointestinal infection ruled out.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms are excluded:

* Gastrointestinal infection or malabsorption.
* Significant acute illness.
* Any identified, untreated cause for failure to thrive other than underlying HIV infection.
* Medical contraindications to megestrol acetate.

Patients with any of the following prior conditions or symptoms are excluded:

Medical contraindications to megestrol acetate including a history of poorly-controlled hypertension, deep venous thrombosis, or heart failure.

History of prior megestrol acetate therapy in the past six months.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Puerto Rico / Med Science Campus, San Juan, Puerto Rico